CLINICAL TRIAL: NCT07028619
Title: Benefits of Bimodal Streaming for MED-EL Cochlear Implants: Early User Experience With the AudioKey Application and Starkey Hearing Aids
Brief Title: Benefits of Bimodal Streaming With MED-EL Cochlear Implants and Starkey Hearing Aids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: US2501
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Sensorineural; Sensorineural Hearing Loss, Bilateral; Cochlear Implant Recipients; Asymmetric Hearing Loss
Keywords: cochlear implants
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Bimodal streaming (Experimental): Bimodal streaming
  Interventions: Device: Bimodal Streaming Configuration

INTERVENTIONS:
Device: Bimodal Streaming Configuration — Participants' devices are configured for bimodal streaming. Participants complete a survey following a trial with the new bimodal streaming feature.

SUMMARY:
This study will evaluate sound quality and user satisfaction with Bluetooth streaming using a new bimodal streaming option for individuals who use a MED-EL cochlear implant and Starkey hearing aid.

DETAILED DESCRIPTION:
MED-EL cochlear implant recipients who use a compatible Starkey hearing aid in the other ear will evaluate a new Bluetooth streaming option that will directly stream audio from their iOS smart device to both hearing devices. A survey will be completed after a trial with the new streaming option.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a MED-EL cochlear implant in one ear
* Using an AudioKey compatible MED-EL audio processor
* Using an AudioKey compatible Starkey hearing aid
* If not using a SONNET 3 audio processor, has access to a MED-EL streaming device
* Using a smartphone that can support the AudioKey application
* Able to complete a survey via cellphone or computer
* Prior experience with Bluetooth streaming or expressed motivation to Bluetooth stream to hearing devices
* Ability to complete all study procedures including provide responses to survey questions

Exclusion Criteria:

* Unable to provide reliable feedback
* Unable to operate a smartphone with or without assistance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-06-26 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Idaho Ear Clinic, Meridian, Idaho, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Bimodal Streaming: Bimodal streaming with DualSync bimodal streaming
Period: Overall Study
Arm/Group | Bimodal Streaming
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bimodal Streaming
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  United States | 10
Duration of Cochlear Implant Experience [Median (Full Range); unit: months] — Months since activation of the cochlear implant
  months | 3.2 [0 to 114.7]

OUTCOME MEASURES:

1. Primary Outcome: User Satisfaction With DualSync Bimodal Streaming Over Existing Bluetooth Streaming Option.
Description: Percentage of participants who reported improvement in subjective listening experience with DualSync bimodal streaming at 1-week. Responses taken from a user survey administered after 1-week with DualSync bimodal streaming.
Time Frame: 1 week
Population: Analysis population differs for questions on streaming music, media, and phone calls as not all participants streamed all forms of audio.
Measure: Count of Participants; unit: Participants
Arm/Group | Bimodal Streaming
Number analyzed (Participants) | 10
Participants
  Participants reporting increased streaming time with DualSync bimodal streaming | 2
  Participants reporting improved clarity with DualSync bimodal streaming | 6
  Participants reporting improved sound quality of music with DualSync bimodal streaming: number analyzed (Participants) | 7
  Participants reporting improved sound quality of music with DualSync bimodal streaming | 7
  Participants reporting increased enjoyment of music with DualSync bimodal streaming: number analyzed (Participants) | 7
  Participants reporting increased enjoyment of music with DualSync bimodal streaming | 6
  Participants reporting improved sound quality of phone calls with DualSync bimodal streaming | 7
  Participants reporting improved ease of listening to phone calls with DualSync bimodal streaming | 7
  Participants reporting improved overall satisfaction with streaming with DualSync bimodal streaming | 6

ADVERSE EVENTS:
Time Frame: From enrollment until completion of 1-week follow-up survey (approximately 1 week)
Arm/Group | Bimodal Streaming
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT07028619/Prot_SAP_000.pdf